CLINICAL TRIAL: NCT00122382
Title: A Phase IIIB Multi-center, Randomized, Double-Blind Study to Evaluate Remission and Joint Damage Progression in Methotrexate Naive Early Erosive RA Subjects Treated With Abatacept Plus Methotrexate Compared With Methotrexate
Brief Title: Remission and Joint Damage Progression in Early Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-023
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Results first posted 2010-07-13 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Rheumatoid Arthritis
Keywords: abatacept, methotrexate, erosive RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABA + MTX (Active Comparator): abatacept 10 mg/kg intravenous (IV) + methotrexate
  Interventions: Drug: Abatacept; Drug: methotrexate
- Placebo (PLA) + MTX (Active Comparator): placebo IV + methotrexate
  Interventions: Drug: Abatacept; Drug: placebo; Drug: methotrexate

INTERVENTIONS:
Drug: Abatacept — abatacept 10 mg/kg IV monthly, methotrexate weekly, for 24 months
Drug: placebo — placebo IV, monthly, methotrexate weekly for 12 months followed by abatacept 10 mg/kg IV monthly, methotrexate weekly for 12 months
  Arms: Placebo (PLA) + MTX
Drug: methotrexate — Oral, titrated to at least 15 mg per week not to exceed 20 mg per week administered every 28 days from Month 12 to Month 24

SUMMARY:
This is a world wide study to evaluate the remission and joint damage in subjects treated with abatacept in addition to methotrexate versus subjects who receive methotrexate along with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) <=2 years; MTX naive or <=10 mg/wk for <=3 weeks. No dose within 3 months prior to informed consent.
* C-Reactive Protein (CRP) >= 4.5 mg/L (after amendment)
* Rheumatoid factor or anti-cyclic citrullinated peptide antibody (anti-CCP) positive
* Tender joints >=12 and swollen joints >=10

Exclusion Criteria:

* Women and men who are not willing to use birth control
* Diagnosed with other rheumatic disease
* History of cancer within 5 years
* Active tuberculosis
* Treatment with another investigation drug within 28 days
* Active bacterial or viral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1052 (Actual)
Dates: Start 2005-07; Primary Completion 2008-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (79):
- United States (19):
  - Rheumatology Associates Of North Alabama, Huntsville, Alabama
  - Talbert Medical Group, Huntington Beach, California
  - Arthritis Assoc And Osteo Ctr Of Col Sprgs, Colorado Springs, Colorado
  - New England Research Associates, Llc, Trumbull, Connecticut
  - Diagnostic Rheumatology And Research, Indianapolis, Indiana
  - Osteoporosis And Clinical Trials Center, Cumberland, Maryland
  - Malamet & Klein, Md, Pa, Hagerstown, Maryland
  - Arthritis Center Of Nebraska, Lincoln, Nebraska
  - Regional Rheumatology Associates, Binghamton, New York
  - Carolina Bone & Joint, Charlotte, North Carolina
  - Physicians East, Pa, Greenville, North Carolina
  - Carolina Pharmaceutical Research, Statesville, North Carolina
  - Lion Research, Norman, Oklahoma
  - Health Research Of Oklahoma, Oklahoma City, Oklahoma
  - Lynn Health Sciences Institute, Oklahoma City, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Low Country Research Center, Charleston, South Carolina
  - Walter F Chase Md Pa, Austin, Texas
  - Arthritis Clinic Of Northern Virginia, P.C., Arlington, Virginia
- Australia (2):
  - Local Institution, Malvern, Victoria
  - Local Institution, Shenton Park, Western Australia
- Belgium (4):
  - Local Institution, Antwerp
  - Local Institution, Brussels
  - Local Institution, Hasselt
  - Local Institution, Leuven
- Brazil (5):
  - Local Institution, Goiânia, Goiás
  - Local Institution, Curitiba, Paraná
  - Local Institution, Rio de Janeiro - Rj, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo, São Paulo
- Canada (7):
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Kitchener, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution, Sherbrooke, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Local Institution, Prague, Czechia
- France (4):
  - Local Institution, Dijon
  - Local Institution, Montpellier
  - Local Institution, Nice
  - Local Institution, Strasbourg
- Germany (3):
  - Local Institution, Berlin
  - Local Institution, Hamburg
  - Local Institution, Leipzig
- Italy (2):
  - Local Institution, Jesi(Ancona)
  - Local Institution, Milan
- Mexico (9):
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, León, Guanajuato
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, D.f., Mexico City
  - Local Institution, Morelia, Michioacan
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, San Luis Potosí City, San Luis Potosí
  - Local Institution, Metepec, State of Mexico
- Netherlands (3):
  - Local Institution, Amsterdam
  - Local Institution, Leiden
  - Local Institution, Nijmegen
- Poland (2):
  - Local Institution, Poznan
  - Local Institution, Warsaw
- Local Institution, Ponce, Puerto Rico
- Local Institution, Moscow, Russia
- South Africa (5):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Muckleneuk, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Berea, KwaZulu-Natal
  - Local Institution, Panorama, Western Cape
- South Korea (4):
  - Local Institution, Anyang
  - Local Institution, Daegu
  - Local Institution, Daejeon
  - Local Institution, Seoul
- Spain (3):
  - Local Institution, A Coruña
  - Local Institution, Santander
  - Local Institution, Seville
- United Kingdom (4):
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Glasgow, Lanarkshire
  - Local Institution, Leeds, North Yorkshire
  - Local Institution, Newcastle, Northumberland

REFERENCES:
- [Derived] Durez P, Westhovens R, Baeke F, Elbez Y, Robert S, Ahmad HA. Identification of poor prognostic joint locations in an early rheumatoid arthritis cohort at risk of rapidly progressing disease: a post-hoc analysis of the Phase III AGREE study. BMC Rheumatol. 2022 Apr 14;6(1):24. doi: 10.1186/s41927-022-00252-4. PMID 35418172
- [Derived] Jansen DTSL, Emery P, Smolen JS, Westhovens R, Le Bars M, Connolly SE, Ye J, Toes REM, Huizinga TWJ. Conversion to seronegative status after abatacept treatment in patients with early and poor prognostic rheumatoid arthritis is associated with better radiographic outcomes and sustained remission: post hoc analysis of the AGREE study. RMD Open. 2018 Mar 30;4(1):e000564. doi: 10.1136/rmdopen-2017-000564. eCollection 2018. PMID 29657830
- [Derived] Smolen JS, Wollenhaupt J, Gomez-Reino JJ, Grassi W, Gaillez C, Poncet C, Le Bars M, Westhovens R. Attainment and characteristics of clinical remission according to the new ACR-EULAR criteria in abatacept-treated patients with early rheumatoid arthritis: new analyses from the Abatacept study to Gauge Remission and joint damage progression in methotrexate (MTX)-naive patients with Early Erosive rheumatoid arthritis (AGREE). Arthritis Res Ther. 2015 Jun 11;17(1):157. doi: 10.1186/s13075-015-0671-9. PMID 26063454
- [Derived] Bathon J, Robles M, Ximenes AC, Nayiager S, Wollenhaupt J, Durez P, Gomez-Reino J, Grassi W, Haraoui B, Shergy W, Park SH, Genant H, Peterfy C, Becker JC, Covucci A, Moniz Reed D, Helfrick R, Westhovens R. Sustained disease remission and inhibition of radiographic progression in methotrexate-naive patients with rheumatoid arthritis and poor prognostic factors treated with abatacept: 2-year outcomes. Ann Rheum Dis. 2011 Nov;70(11):1949-56. doi: 10.1136/ard.2010.145268. Epub 2011 Aug 6. PMID 21821865

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1052 participants were enrolled, 541 were not randomized (2 for adverse events, 32 subjects withdrew consent, 1 pregnancy, 6 lost to follow-up, 470 no longer met study criteria, 30 for other reasons).
Groups:
- Abatacept (ABA) + Methotrexate (MTX) (Double-Blind): ABA 10 mg/kg (weight-tiered dose) intravenous (IV) infusions in combination with oral MTX titrated to at least 15 mg per week not to exceed 20 mg per week. Study drug administered on Days 1, 15, 29 and every 28 days thereafter up to Month 12 (end of double blind period).
- Placebo (PLA) + Methotrexate (MTX) (Double-Blind): Placebo (Dextrose 5% Water for Injection U.S.P. [D5W] or Normal Saline [NS] IV infusions in combination with oral MTX) titrated to at least 15 mg per week not to exceed 20 mg per week. Administered on Days 1, 15, 29, and every 28 days thereafter up to Month 12 (end of double blind period).
- ABA + MTX (Open-Label): Participants who received ABA + MTX in the 12-month, open-label period of the study (including 232 subjects who previously received ABA + MTX and 227 subjects who previously received PLA + MTX in the 12-month, double-blind period of the study). ABA 10 mg/kg (weight-tiered dose) intravenous (IV) infusions in combination with weekly oral MTX were administered every 28 days from Month 12 to Month 24 (open-label period).
Period: Double-Blind Study
Arm/Group | Abatacept (ABA) + Methotrexate (MTX) (Double-Blind) | Placebo (PLA) + Methotrexate (MTX) (Double-Blind) | ABA + MTX (Open-Label)
Started | 256 (participants randomized) | 255 (participants randomized) | 0
Treated | 256 | 253 | 0
Completed | 232 | 227 | 0
Not Completed | 24 | 28 | 0
Not completed — Adverse Event | 9 | 11 | 0
Not completed — Death | 2 | 2 | 0
Not completed — Lack of Efficacy | 0 | 8 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Pregnancy | 2 | 0 | 0
Not completed — Subject No Longer Meets Study Criteria | 1 | 0 | 0
Not completed — Withdrawal of Consent | 7 | 3 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Methotrexate Discontinued | 0 | 1 | 0
Not completed — Randomized but not treated | 0 | 2 | 0
Period: Open-Label Study
Arm/Group | Abatacept (ABA) + Methotrexate (MTX) (Double-Blind) | Placebo (PLA) + Methotrexate (MTX) (Double-Blind) | ABA + MTX (Open-Label)
Started | 0 | 0 | 459
Completed | 0 | 0 | 433
Not Completed | 0 | 0 | 26
Not completed — Adverse Event | 0 | 0 | 11
Not completed — Death | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Pregnancy | 0 | 0 | 2
Not completed — Poor/Non-Compliance | 0 | 0 | 1
Not completed — Withdrawal of Consent | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- ABA + MTX (Double-Blind): ABA 10 mg/kg (weight-tiered dose) intravenous (IV) infusions in combination with oral MTX titrated to at least 15 mg per week not to exceed 20 mg per week. Study drug administered on Days 1, 15, 29 and every 28 days thereafter up to Month 12.
- PLA + MTX (Double-Blind): Placebo (Dextrose 5% Water for Injection U.S.P. [D5W] or Normal Saline [NS] IV infusions in combination with oral MTX titrated to at least 15 mg per week not to exceed 20 mg per week. Administered on Days 1, 15, 29, and every 28 days thereafter up to Month 12.
- Total: Total of all reporting groups
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind) | Total
Number analyzed (Participants) | 256 | 253 | 509
Age Continuous [Mean (Standard Deviation); unit: years] | 50.1 (12.4) | 49.7 (13.0) | 49.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 199 | 395
  Male | 60 | 54 | 114
Anti-Cyclic Citrullinated Peptide 2 (CCP2) Status [Number; unit: participants] — Anti-CCP2 antibodies are autoantibodies that react with citrullinated proteins, are frequent in Rheumatoid Arthritis and are associated with erosive disease. > 5 units/mL is a positive result.
  participants
    unknown | 2 | 0 | 2
    positive | 236 | 217 | 453
    negative | 18 | 36 | 54
Duration of Rheumatoid Arthritis (RA) Disease [Number; unit: participants]
  </= 6 months | 167 | 157 | 324
  > 6 months - 12 months | 36 | 34 | 70
  > 12 months | 53 | 62 | 115
Rheumatoid Factor (RF) Status [Number; unit: participants] — Rheumatoid Factor is an autoantibody that is usually present in the serum of people with rheumatoid arthritis. The cut-point value for seroconversion was 15 IU/mL (>/= 15 IU/mL resulted in a positive result).
  participants
    unknown | 1 | 1 | 2
    positive | 246 | 245 | 491
    negative | 9 | 7 | 16
Disease Activity Scale 28 (DAS 28) C-reactive Protein (CRP) [Mean (Standard Deviation); unit: units on a scale] — DAS 28-CRP=continuous composite of 4 variables: number of tender joints out of 28, number of swollen joints out of 28, CRP in milligrams/Liter (mg/L), and subject assessment of disease activity measured on a Visual Analogue Scale (VAS) of 100 millimeters (mm). Current disease activity is presented on a scale of 0 to 10, with a score above 5.1=high disease activity and below 3.2=low disease activity. VAS=a measurement instrument for characteristics that range across a continuum of values. Range is 1 to 100; a lower value signifies improvement. 1 participant in Placebo group was not evaluated.
  units on a scale | 6.3 (1.0) | 6.2 (1.0) | 6.3 (1.0)
Duration of RA [Mean (Standard Deviation); unit: months] | 6.2 (7.5) | 6.7 (7.1) | 6.5 (7.3)
Erosion Score [Mean (Standard Deviation); unit: units on a scale] — To assess joint damage progression, the Genant-modified Sharp scoring method was used to evaluate radiographs of hands/wrists and feet for erosions and JSN. The erosion score range is 0 (no radiographic damage) to 145 (worst possible radiographic damage). Higher scores indicated more damage. 3 participants in the abatacept group were not included in the measure.
  units on a scale | 5.4 (6.1) | 4.8 (5.4) | 5.1 (5.8)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — HAQ-DI=self-reported measure of physical function calculated as a mean of 8 category scores: Dressing/Grooming, Rising, Eating, Walking, Hygiene, Reach, Grip, Activities. Each category score is calculated as the maximum of the scores for the questions within the category. HAQ-DI is expressed on a scale of 0 (without any difficulty) to 3 (unable to do) representing an average score across the category. Scores for at least 6 categories are needed to compute HAQ score. Changes to lower scores=improvement in physical function. 2 participants in the abatacept and placebo groups were not evaluated.
  units on a scale | 1.7 (0.7) | 1.7 (0.7) | 1.7 (0.7)
Joint Space Narrowing (JSN) Score [Mean (Standard Deviation); unit: units on a scale] — To assess joint damage progression, the Genant-modified Sharp scoring method was used to evaluate radiographs of hands/wrists and feet for erosions and JSN. The joint space narrowing score range is 0 (no radiographic damage) to 145 (worst possible radiographic damage). Higher scores indicated more damage. 3 participants in the abatacept group were not included in the measure.
  units on a scale | 2.1 (4.2) | 1.9 (4.0) | 2.0 (4.1)
Physician Global Assessment per Visual Analogue Scale (VAS) [Mean (Standard Deviation); unit: mm] — Physician Global Assessment is measured by VAS (100 mm). A Visual Analogue Scale (VAS) is a measurement instrument for characteristics that range across a continuum of values. Range is 1-100; a lower score indicates a better Physician Assessment of Global Health. 1 participant in the abatacept group was not evaluated for this measure.
  mm | 67.1 (18.2) | 65.7 (18.9) | 66.4 (18.5)
Subject Global Assessment per VAS [Mean (Standard Deviation); unit: mm] — Subject Global Assessment is measured by VAS (100 mm). A Visual Analogue Scale (VAS) is a measurement instrument for characteristics that range across a continuum of values. Range is 1-100; a lower score indicates a better Subject Assessment of Global Health. 1 participant in the Placebo group was not evaluated for this measure.
  mm | 65.8 (21.8) | 63.7 (24.0) | 64.8 (22.9)
Subject Pain Assessment per VAS [Mean (Standard Deviation); unit: mm] — Subject Pain Assessment measured by VAS (100 mm). A Visual Analogue Scale (VAS) is a measurement instrument for characteristics that range across a continuum of values. Range is 1-100; a lower value signifies a better subject pain assessment. 1 participant in the Placebo group was not evaluated for this measure.
  mm | 66.6 (22.5) | 67.1 (22.6) | 66.8 (22.5)
Swollen Joints [Mean (Standard Deviation); unit: number of swollen joints] — Total number of joints analyzed=66
  number of swollen joints | 22.9 (11.3) | 21.9 (10.1) | 22.4 (10.8)
Tender Joints [Mean (Standard Deviation); unit: number of tender joints] — Total number of joints analyzed=68
  number of tender joints | 31.3 (14.8) | 30.8 (14.0) | 31.0 (14.4)
Total Genant-modified Sharp score [Mean (Standard Deviation); unit: units on a scale] — To assess joint damage progression, the Genant-modified Sharp scoring method was used to evaluate radiographs of hands/wrists and feet for erosions and JSN. The total Genant-modified Sharp score ranges from 0 (no radiographic damage) to 290 (worst possible radiographic damage) and is the sum of the erosion score (range 0-145) and the joint space narrowing score (range 0-145). Higher scores indicated more damage. 3 participants in the abatacept group were not included in the measure.
  units on a scale | 7.5 (9.7) | 6.7 (8.8) | 7.1 (9.2)

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With American College of Rheumatology (ACR) 50 Response at Month 12
Description: ACR 50 response was defined as a 50% improvement from baseline to Month 12 in tender and swollen joint counts and 50% improvement in 3 of the remaining 5 core set measures (subject global assessment of pain, subject global assessment of disease activity, physician global assessment of disease activity, subject assessment of physical function), and 1 acute phase reactant value [ie, CRP].
Time Frame: Month 12
Population: Intention-to-Treat=All randomized and treated; all missing data subsequent to discontinuation are considered non-responders.
Measure: Number; unit: participants
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 256 | 253
participants | 147 | 107
Statistical Analysis 1: Comparison: ABA + MTX (Double-Blind) vs PLA + MTX (Double-Blind); Estimated Difference between ABA and PLA is the estimated difference between ABA and PLA in the proportion of subjects achieving an ACR 50 response; Test type: Superiority or Other; p < 0.001, Chi-squared, Continuity-Corrected — p-value of <0.05: probability for testing the difference between ABA and PLA; Estimated Difference between ABA and PLA = 15.1, 95% CI 2-sided [6.0 to 24.2]

2. Secondary Outcome: Number of Participants With Major Clinical Response (MCR) at Month 12
Description: MCR was defined as 6 months of consecutive ACR 70 response at Month 12. ACR 70, the American College of Rheumatology (ACR) definition of 70% improvement was based on a 70% improvement (compared to baseline values) in tender and swollen joint counts and 70% improvement in 3 of the remaining 5 core set measures (subject global assessment of pain, subject global assessment of disease activity, physician global assessment of disease activity, subject assessment of physical function, and 1 acute phase reactant value [ie, CRP]).
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 256 | 253
participants | 70 | 30
Statistical Analysis 1: Comparison: ABA + MTX (Double-Blind) vs PLA + MTX (Double-Blind); Estimated Difference between ABA and PLA is the estimated difference between ABA and PLA in the proportion of subjects achieving MCR; Test type: Superiority or Other; p < 0.001, Chi-squared, Continuity-Corrected — p-value of <0.05: probability for testing the difference between ABA and PLA; Estimated Difference between ABA and PLA = 15.5, 95% CI 2-sided [8.2 to 22.8]

3. Secondary Outcome: Adjusted Mean Change From Baseline in DAS-28-CRP Score to Month 12
Description: DAS 28-CRP is a continuous variable that is a composite of 4 variables: the number of tender joints out of 28 joints, the number of swollen joints out of 28 joints, CRP in milligrams/Liter (mg/L), and subject assessment of disease activity measure on a Visual Analogue Scale (VAS) of 100 millimeters (mm). The DAS28 scale=0 to 10, indicating the current activity of the rheumatoid arthritis. A DAS28 >5.1=high disease activity; <3.2=low disease activity; <2.6=remission. Change from Baseline=Post-baseline - Baseline value; Adjusted for baseline value.
Time Frame: Baseline, Month 12
Population: Last Observation Carried Forward (LOCF) Intent to Treat population = all randomized and treated. As change from baseline analysis, only those with baseline and post-baseline included.
Measure: Mean (Standard Error); unit: units in a scale
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 253 | 251
units in a scale | -3.22 (0.09) | -2.49 (0.09)
Statistical Analysis 1: Comparison: ABA + MTX (Double-Blind) vs PLA + MTX (Double-Blind); Test type: Superiority or Other; p < 0.001, ANCOVA — p-value of <0.05: probability for testing the difference between ABA and PLA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Estimate of/Adjusted Difference = -0.73, 95% CI 2-sided [-0.98 to -0.48]

4. Secondary Outcome: Number of Participants With Health Assessment Questionnaire (HAQ) Response at Month 12
Description: Physical function was evaluated using the HAQ-disability index (HAQ-DI), a questionnaire with 20 questions assessing function in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and common activities. The questions are evaluated on a 4-point scale: 0 = without any difficulty; 1 = with some difficulty; 2 = with much difficulty; 3 = unable to do. The 8 category scores are averaged into an overall HAQ-DI score on a scale from 0 (no disability) to 3 (completely disabled). Higher scores indicate greater dysfunction. HAQ response=improvement of at least 0.3 units from baseline.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 256 | 253
participants | 184 | 157
Statistical Analysis 1: Comparison: ABA + MTX (Double-Blind) vs PLA + MTX (Double-Blind); Estimated Difference between ABA and PLA is the estimated difference between ABA and PLA in the proportion of subjects achieving HAQ response; Test type: Superiority or Other; p = 0.024, Chi-squared, Continuity-Corrected — p-value of <0.05: probability for testing the difference between ABA and PLA; Estimated Difference between ABA and PLA = 9.8, 95% CI 2-sided [1.3 to 18.4]

5. Secondary Outcome: Adjusted Mean Change in Short Form 36 (SF-36) From Baseline to Month 12
Description: The SF-36 covers 8 health dimensions: 4 physical subscales (physical function, role-physical, bodily pain, and general health) and 4 mental subscales (vitality, social function, role-emotional, and mental health). The scores range from 0 to 100, with a higher score indicating better quality of life. Two summary scores (physical and mental component summaries) were produced taking a weighted linear combination of the 8 individual subscales. Change from Baseline=Post-baseline - Baseline value; adjusted for baseline value.
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 254 | 249
units on a scale
  Physical Component Summary (PCS) Score | 11.68 (0.62) | 9.18 (0.63)
  Mental Component Summary (MCS) Score | 8.15 (0.64) | 6.34 (0.64)
Statistical Analysis 1: Comparison: ABA + MTX (Double-Blind) vs PLA + MTX (Double-Blind); PCS Adjusted Mean Change from Baseline to Month 12; Test type: Superiority or Other; p = 0.005, ANCOVA — p-value of <0.05: probability for testing the difference between ABA and PLA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Estimate of/Adjusted Difference = 2.50, 95% CI 2-sided [0.77 to 4.23]
Statistical Analysis 2: Comparison: ABA + MTX (Double-Blind) vs PLA + MTX (Double-Blind); MCS Adjusted Mean Change from Baseline to Month 12; Test type: Superiority or Other; p = 0.046, ANCOVA — p-value of <0.05: probability for testing the difference between ABA and PLA; Adjustment based on ANCOVA model with treatment as factor and baseline value as covariate; Estimate of/Adjusted Difference = 1.81, 95% CI 2-sided [0.03 to 3.60]

6. Secondary Outcome: Mean Change From Baseline in Radiographic Erosion and Joint Space Narrowing (JSN) Scores to Month 12
Description: To assess joint damage progression, the Genant-modified Sharp scoring method was used to evaluate radiographs of hands/wrists and feet for erosions and JSN. The erosion score range is 0 (no radiographic damage) to 145 (worst possible radiographic damage). The joint space narrowing score range is 0 (no radiographic damage) to 145 (worst possible radiographic damage). Higher scores indicated more damage. Change from baseline = Post-baseline - Baseline value
Time Frame: Baseline, Month 12
Population: Intention-to-Treat - linear extrapolation imputation. Analysis of change from baseline restricts subjects included in to the analysis to those with baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 242 | 242
units on a scale
  Baseline Mean Erosion Score | 5.48 (6.15) | 4.81 (5.46)
  Mean Change from Baseline in Erosion Score | 0.50 (1.39) | 0.89 (2.24)
  Baseline Mean JSN Score | 2.03 (3.99) | 1.86 (3.95)
  Mean Change from Baseline in JSN Score | 0.13 (0.53) | 0.17 (0.54)
Statistical Analysis 1: Comparison: ABA + MTX (Double-Blind) vs PLA + MTX (Double-Blind); comparison of change in erosion scores between abatacept and placebo; Test type: Superiority or Other; p = 0.033, Nonparametric ANCOVA — P-value of <0.05: probability for comparison of change in radiographic scores between abatacept and placebo
Statistical Analysis 2: Comparison: ABA + MTX (Double-Blind) vs PLA + MTX (Double-Blind); comparison of change in JSN scores between abatacept and placebo; Test type: Superiority or Other; p = 0.353, Nonparametric ANCOVA — P-value of <0.05: probability for comparison of change in radiographic scores between abatacept and placebo

7. Secondary Outcome: Number of Participants With Anti-abatacept or Anti-CTLA4-T Responses in the Double-blind Period as Analyzed by Enzyme-linked-immunosorbent Serologic Assay (ELISA)
Description: Serum samples were analyzed by ELISA to detect antibodies against the whole molecule (both CTLA4 and Ig [anti-abatacept antibody]) or solely to CTLA4 (anti-CTLA4-T antibody). Reported as titer, the reciprocal of the sample dilution which yielded a signal equivalent to the statistically set cut point for the assay. For the anti-abatacept assay, minimum required dilution is 400-fold, therefore seronegative samples are those < lowest reportable titer (<400). For the anti-CTLA4-T assay, minimum required dilution is 25-fold, therefore seronegative samples are those < lowest reportable titer (<25).
Time Frame: includes data up to approximately 85 days past the last dose of the double-blind period or start of the open-label period, whichever occurred first.
Population: Treated participants in the double-blind period who were evaluated for anti-abatacept or anti-CTLA4-T responses
Measure: Number; unit: Participants
Groups:
- ABA+ MTX On-treatment; ABA + MTX Post-discontinuation: ABA 10 mg/kg (weight-tiered dose) intravenous (IV) infusions in combination with oral MTX titrated to at least 15 mg per week not to exceed 20 mg per week. Study drug administered on Days 1, 15, 29 and every 28 days thereafter up to Month 12.
Arm/Group | ABA+ MTX On-treatment | ABA + MTX Post-discontinuation
Number analyzed (Participants) | 249 | 13
Participants
  Anti-abatacept Responses | 3 | 0
  Anti-CTLA4-T Responses | 1 | 1

8. Primary Outcome: Number of Participants in DAS 28 C-reactive Protein (CRP) Remission at Month 12
Description: Number of participants who achieved remission at Month 12 of treatment, as defined by a Disease Activity Score (DAS) 28-CRP score of <2.6. DAS 28-CRP is a continuous measure, a composite of 4 variables: number of tender joints out of 28 joints, number of swollen joints out of 28 joints, CRP (in mg/L), and subject assessment of disease activity measure on a Visual Analogue Scale (VAS) of 100 millimeters (mm). The DAS28 scale=0 (best) to 10 (worst), indicating the current activity of the rheumatoid arthritis. A DAS28 >5.1 = high disease activity; <=3.2 = low disease activity; <2.6 = remission.
Time Frame: Month 12
Population: Intent to treat = all randomized and treated subjects. Those with missing data post-discontinuation were considered non-responders.
Measure: Number; unit: participants
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 256 | 253
participants | 106 | 59
Statistical Analysis 1: Comparison: ABA + MTX (Double-Blind) vs PLA + MTX (Double-Blind); Estimated Difference between ABA and PLA is the estimated difference between ABA and PLA in the proportion of subjects achieving DAS28-CRP remission; Test type: Superiority or Other; p < 0.001, Chi-squared, Continuity-Corrected — Total score was tested only if there was statistical significance in remission rate. For each test, the nominal type I error rate is set at 5%; this sequential testing procedure preserves the overall type I error rate at 5%; Estimated Difference between ABA and PLA = 18.1, 95% CI 2-sided [9.6 to 26.6]

9. Primary Outcome: Mean Change From Baseline in Radiographic Total Score to Month 12
Description: To assess joint damage progression, the Genant-modified Sharp scoring method was used to evaluate radiographs of hands/wrists and feet for erosions and joint space narrowing (JSN). The total Genant-modified Sharp score ranges from 0 (no radiographic damage) to 290 (worst possible radiographic damage) and is the sum of the erosion score (range 0-145) and the joint space narrowing score (range 0-145). Higher scores indicated more damage.
Time Frame: Baseline, Month 12
Population: The analysis was intent-to-treat. Because the analysis was change from baseline, only those with baseline and post-baseline were included. Linear extrapolation imputation was applied.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 242 | 242
units on a scale
  Baseline Mean | 7.50 (9.52) | 6.67 (8.71)
  Mean Change from Baseline | 0.63 (1.74) | 1.06 (2.45)
Statistical Analysis 1: Comparison: ABA + MTX (Double-Blind) vs PLA + MTX (Double-Blind); Test type: Superiority or Other; p < 0.040, non-parametric ANCOVA — [p-value comment as in outcome 8, analysis 1]

10. Primary Outcome: Number of Subjects With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, and Discontinuations Due to AEs During the Open-Label Period
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. Related AE/SAE=Certain, Probable, Possible, or Missing. SAE=any untoward medical occurrence that results in death, is life-threatening, requires or prolongs inpatient hospitalization (including elective surgery), results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: Continuously through open-label period (from Month 12 to Month 24). Includes data up to 56 days post last dose in the open-label period or start of the maintenance sub-study, whichever occurred first.
Population: All subjects who received at least 1 dose of ABA in the open-label period were included in the safety analyses.
Measure: Number; unit: participants
Groups:
- ABA + MTX (Open-Label): Participants who received ABA + MTX in the 12-month, open-label period of the study (including 232 subjects who previously received ABA + MTX and 227 subjects who previously received PLA + MTX in the 12-month, double-blind period of the study). ABA 10 mg/kg (weight-tiered dose) intravenous (IV) infusions in combination with oral MTX titrated to at least 15 mg per week not to exceed 20 mg per week was administered every 28 days from Month 12 to Month 24 (open-label period).
Arm/Group | ABA + MTX (Open-Label)
Number analyzed (Participants) | 459
participants
  AEs | 345
  Related AEs | 128
  SAEs | 29
  Related SAEs | 10
  Discontinuations due to AEs | 11
  Discontinuations due to SAEs | 4
  Deaths | 2

11. Primary Outcome: Number of Participants With Serious Adverse Events Reported During the Open-Label Period
Description: SAE=any untoward medical occurrence that results in death, is life-threatening, requires or prolongs inpatient hospitalization (including elective surgery), results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: as for outcome 10
Population: All subjects who received at least 1 dose of ABA in the open-label period were included in the safety analyses.
Measure: Number; unit: participants
Groups:
- ABA + MTX (Open Label): Participants who received ABA + MTX in the 12-month, open-label period of the study (including 232 subjects who previously received ABA + MTX and 227 subjects who previously received PLA + MTX in the 12-month, double-blind period of the study). ABA 10 mg/kg (weight-tiered dose) intravenous (IV) infusions in combination with oral MTX titrated to at least 15 mg per week not to exceed 20 mg per week was administered every 28 days from Month 12 to Month 24 (open-label period).
Arm/Group | ABA + MTX (Open Label)
Number analyzed (Participants) | 459
participants
  Any SAE | 29
  Infections and infestations | 8
  Gastrointestinal disorders | 4
  Nervous system disorders | 4
  Cardiac disorders | 3
  Hepatobiliary disorders | 3
  Eye disorders | 2
  Musculoskeletal and connective tissue disorders | 2
  Vascular disorders | 2
  Immune System Disorders | 1
  Injury, Poisoning, and Procedural Complications | 1
  Investigations | 1
  Metabolism and Nutrition Disorders | 1
  Renal and Urinary Disorders | 1
  Respiratory, Thoracic, and Mediastinal Disorders | 1

12. Secondary Outcome: Number of Participants With Anti-abatacept or Anti-CTLA4-T Responses During the Open-Label Period (From Month 12 to Month 24) as Analyzed by ELISA
Description: as for outcome 7
Time Frame: Includes open-label data up to approximately 85 days post last dose in the open-label period or start of the maintenance sub-study, whichever occurred first.
Population: Treated participants in the open-label period were evaluated for anti-abatacept or anti-CTLA4-T responses
Measure: Number; unit: participants
Arm/Group | Anti-Abatacept Antibody Response | Anti-CTLA4-T Antibody Response
Number analyzed (Participants) | 451 | 456
participants | 13 | 16

13. Secondary Outcome: Number of Participants With Health Assessment Questionnaire (HAQ) Response at Month 24
Description: as for outcome 4
Time Frame: Baseline, Month 24
Population: All treated participants in the Open-label period. Treatment groups represent treatment received in the Double Blind Period.
Measure: Number; unit: participants
Groups:
- ABA + MTX (Double-Blind); PLA + MTX (Double-Blind): Participants who received ABA + MTX in the 12-month, open-label period of the study (including 232 subjects who previously received ABA + MTX and 227 subjects who previously received PLA + MTX in the 12-month, double-blind period of the study). ABA 10 mg/kg (weight-tiered dose) intravenous (IV) infusions in combination with oral MTX titrated to at least 15 mg per week not to exceed 20 mg per week was administered every 28 days from Month 12 to Month 24 (open-label period). The groups are determined by treatment status in the double blind period to observe efficacy differences.
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 232 | 227
participants | 189 | 178

14. Secondary Outcome: Mean Change From Baseline in Radiographic Total, Erosion and JSN Scores to Month 24
Description: To assess joint damage progression, the Genant-modified Sharp scoring method was used to evaluate radiographs of hands/wrists and feet for erosions and JSN. The total Genant-modified Sharp score ranges from 0 (no radiographic damage) to 290 (worst possible radiographic damage) and is the sum of the erosion score (range 0-145) and the joint space narrowing score (range 0-145). Higher scores indicated more damage. Change from baseline = Postbaseline - baseline value.
Time Frame: Baseline, Month 24
Population: All treated participants in the open-label period. Because the analysis was change from baseline, only those with baseline and post-baseline were included. Linear extrapolation imputation was applied. Treatment groups represent treatment received in the double-blind period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 213 | 192
units on a scale
  Erosion Score Baseline Mean | 5.91 (6.48) | 5.49 (5.85)
  Erosion Score Mean Change from Baseline | 0.59 (2.31) | 1.40 (3.08)
  JSN Score Baseline Mean | 1.83 (3.82) | 1.75 (3.92)
  JSN Score Mean Change from Baseline | 0.25 (1.03) | 0.34 (0.99)
  Total Score Baseline Mean | 7.73 (9.50) | 7.24 (8.89)
  Total Score Mean Change from Baseline | 0.84 (3.22) | 1.75 (3.59)

15. Primary Outcome: Number of Participants With SAEs With an Outcome of Death During the Open-label Period
Description: Any untoward medical occurrence (SAE) that resulted in death
Time Frame: as for outcome 10
Population: All subjects who received at least 1 dose of ABA in the open-label period were included in the safety analyses.
Measure: Number; unit: participants
Arm/Group | ABA + MTX (Open-Label)
Number analyzed (Participants) | 459
participants
  Pneumonia | 1
  Pneumonia/septic shock | 1

16. Primary Outcome: Incidence Rates of Autoimmune Disorders in ABA-Treated Participants
Description: The incidence rates of autoimmune disorders are defined as the (number of patients experiencing the event/exposure within the period)*100 and are expressed in 100 person-years. Subjects experiencing the event had their exposure censored at the time of the 1st event.
Time Frame: Double Blind Period (+56 days post last dose in double-blind period or start of open-label period, whichever came first). Open-label period (56 days post last dose in the open-label period or start of maintenance sub-study, whichever came first).
Population: All subjects who received at least 1 dose of abatacept. Double-blind (DB) period: all treated in DB period; Open-label (OL) Period: all treated in OL period.
Measure: Number; unit: Number of participants/100 patient-years
Arm/Group | ABA + MTX (Double-Blind) | ABA + MTX (Open-Label)
Number analyzed (Participants) | 256 | 459
Number of participants/100 patient-years | 2.47 | 1.30

17. Primary Outcome: Incidence Rates of Infections and Infestations of Adverse Events in ABA-Treated Participants
Description: The incidence rates of infections and infestations are defined as the (number of patients experiencing the event /exposure within the period)*100 and are expressed in 100 person-years. Subjects experiencing the event had their exposure censored at the time of the 1st event.
Time Frame: Double Blind Period (+56 days post last dose in double-blind period or start of the open-label period, whichever came first). Open-label period (56 days post last dose in open-label period or start of maintenance sub-study, whichever came first).
Population: as for outcome 16
Measure: Number; unit: Number of patients/100 patient-years
Arm/Group | ABA + MTX (Double-Blind) | ABA + MTX (Open-Label)
Number analyzed (Participants) | 256 | 459
Number of patients/100 patient-years | 78.37 | 66.68

18. Primary Outcome: Incidence Rates of Malignant Neoplasm Adverse Events in ABA-Treated Participants
Description: The incidence rates of malignant neoplasms are defined as the (number of patients experiencing the event /exposure within the period)*100 and are expressed in 100 person-years. Subjects experiencing the event had their exposure censored at the time of the 1st event.
Time Frame: as for outcome 17
Population: as for outcome 16
Measure: Number; unit: number of patients/100 patient-years
Arm/Group | ABA + MTX (Double-Blind) | ABA + MTX (Open-Label)
Number analyzed (Participants) | 256 | 459
number of patients/100 patient-years | 0.81 | 0

19. Primary Outcome: Number of Participants With a Serious Acute-Infusional AE of Anaphylactic Shock During Open-Label Period
Description: There were 107 Prespecified, acute-infusional SAEs (occurring within 1 hour after the start of study drug infusion) pre-specified in the protocol; anaphylactic shock was the only one occuring in this study.
Time Frame: Open-Label Period (Month 12 to Month 24)
Population: All participants treated during the Open-Label period.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX (Open-label)
Number analyzed (Participants) | 459
Participants | 1

20. Primary Outcome: Number of Participants With Select Blood Chemistry Laboratory Values Meeting the Marked Abnormality Criteria During the Open-Label Period
Description: Number of subjects with high liver function and kinedy tests: alkaline phosphatase (ALP) >2x upper limit of normal (ULN) or if pretreatment (PRE-RX) >ULN then >3x PRE-RX; aspartate aminotransferase (AST) >3x ULN or if PRE-RX >ULN then >4x PRE-RX; alanine aminotransferase (ALT) >3x ULN or if PRE-RX >ULN then >4x PRE-RX; g-glutamyl transferase (GGT)>2x ULN or if PRE-RX >ULN then >3x PRE-RX; total bilirubin >2x ULN or if PRE-RX >ULN then >4x PRE-RX; blood urea nitrogen >2x PRE-RX; creatinine >1.5x PRE-RX.
Time Frame: as for outcome 10
Population: All Treated participants in the Open-label Period; n=number of participants evaluated for this measure.
Measure: Number; unit: participants
Arm/Group | ABA + MTX (Open-Label)
Number analyzed (Participants) | 459
participants
  ALP (n=459) | 2
  AST (n=459) | 10
  ALT (n=459) | 24
  GGT (n=459) | 15
  Total Bilirubin (n=459) | 0
  Blood Urea Nitrogen (n=459) | 13
  Creatinine (n=457) | 81

21. Primary Outcome: Number of Participants With Hematology Laboratory Values Meeting the Marked Abnormality Criteria During the Open-Label Period
Description: Marked abnormalities in hemoglobin >3 g/dL decrease from PRE-RX; hematocrit <0.75x PRE-RX; erythrocytes <0.75x PRE-RX; platelet count <0.67x lower limit of normal (LLN) or >1.5x ULN or if PRE-RX <LLN then <0.5x PRE-RX and <100,000/mm3; leukocytes <0.75x LLN or >1.25x ULN or if PRE-RX <LLN then <0.8x PRE-RX or >ULN if PRE-RX >ULN then >1.2x PRE-RX or <LLN; neutrophils if value <1.00 x10^3 c/uL; lymphocytes if value <.750 x10^3 c/uL or if value >7.50 x10^3 c/uL; monocytes if value >2000/MM3; basophils if value >400/mm3; eosinophils if value >.750 x10^3 c/uL
Time Frame: Continuously from start of open-label period up to 56 days post the last dose in the open-label period or start of the maintenance sub-study, whichever occurred first.
Population: All participants treated during the open-label period; n= number of participants evaluated for this measure.
Measure: Number; unit: participants
Arm/Group | ABA + MTX (Open-Label)
Number analyzed (Participants) | 459
participants
  Low Hemoglobin (n=458) | 9
  Low Hematocrit (n=458) | 5
  Low Erythrocyte (n=458) | 8
  Low Platelet Count (n=455) | 1
  High Platelet Count (n=455) | 1
  Low Leukocytes (n=458) | 14
  High Leukocytes (n=458) | 12
  Low Neutrophils + Bands (absolute) (n=459) | 6
  Low Lymphocytes (absolute) (n=459) | 39
  High Lymphocytes (absolute) (n=459) | 1
  High Monocytes (absolute) (n=459) | 0
  High Basophils (absolute) (n=459) | 2
  High Eosinophils (absolute) (n=459) | 19

22. Secondary Outcome: Number of Participants Without Radiographic Progression (as Measured by in Erosion Scores, JSN Scores, and Total Scores) From Baseline at Month 24
Description: Participants with no radiographic progression (defined as change in score <=0 or <=0.5), from baseline to Month 24. To assess joint damage progression, the Genant-modified Sharp scoring method was used to evaluate radiographs of hands/wrists and feet for erosions and JSN. The total Genant-modified Sharp score ranges from 0 (no radiographic damage) to 290 (worst possible radiographic damage) and is the sum of the erosion score (range 0-145) and the joint space narrowing score (range 0-145). Higher scores indicated more damage.
Time Frame: Baseline, Month 24
Population: All treated participants in the open-label period. Treatment groups represent treatment received in the double-blind period.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 213 | 192
Participants
  Change from Baseline <= 0 in Erosion Score | 125 | 92
  Change from Baseline <= 0.5 in Erosion Score | 144 | 114
  Change from Baseline <= 0 in JSN Score | 175 | 150
  Change from Baseline <= 0.5 in JSN Score | 190 | 166
  Change from Baseline <= 0 in Total Score | 121 | 84
  Change from Baseline <= 0.5 in Total Score | 139 | 107

23. Secondary Outcome: Number of Participants Without Radiographic Progression (as Measured by in Erosion Scores, JSN Scores, and Total Scores) at Month 24 in Participants Without Progression at Month 12
Description: Participants with no radiographic progression ((defined as change in score <=0 or <=0.5), sustained from Month 12 and Month 24. To assess joint damage progression, the Genant-modified Sharp scoring method was used to evaluate radiographs of hands/wrists and feet for erosions and JSN. The total Genant-modified Sharp score ranges from 0 (no radiographic damage) to 290 (worst possible radiographic damage) and is the sum of the erosion score (range 0-145) and the joint space narrowing score (range 0-145). Higher scores indicated more damage.
Time Frame: Month 12, Month 24
Population: Number of Participants Analyzed=All treated participants in the open-label period. (Treatment groups represent treatment received in the double-blind period.) n=the number of subjects with observed data included in the analysis.
Measure: Number; unit: Participants
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 232 | 227
Participants
  Erosion Score Sustained <=0 (n=125; n=100) | 116 | 87
  Erosion Score Sustained <=0.5 (n=145; n=114) | 135 | 107
  JSN Score Sustained <=0 (n=180; n=165) | 169 | 150
  JSN Score Sustained <=0.5 (n=192; n=177) | 185 | 163
  Total Score sustained <=0 (n=123; n=97) | 112 | 81
  Total Score sustained <=0.5 (n=144; n=112) | 131 | 101

24. Secondary Outcome: Mean Difference Observed in Change From Baseline to Month 12 and Between Month 12 and Month 24 in Radiographic Scores (Total Score)
Description: Mean difference observed in change from baseline to Month 12 and between Month 12 and Month 24 in radiographic scores (Total Score). To assess joint damage, the Genant-modified Sharp scoring method was used to evaluate radiographs of hands/wrists and feet for erosions and JSN. The total Genant-modified Sharp score ranges from 0 (no radiographic damage) to 290 (worst possible radiographic damage) and is the sum of the erosion score (range 0-145) and the joint space narrowing score (range 0-145). Higher scores indicated more damage.
Time Frame: Baseline, Month 12, Month 24
Population: Analysis includes all treated participants in the open-label period originally randomized to abatacept. Analysis includes all participants with observed assessments collected at Baseline (Day 1), Day 365 (Month 12), and Day 729 (Month 24)
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Year 1 Change: Year 1 Change = Day 365 - Day 1
- Year 2 Change: Year 2 Change = Day 729 (Month 24) - Day 365 (Month 12)
Arm/Group | Year 1 Change | Year 2 Change
Number analyzed (Participants) | 207 | 207
units on a scale | 0.66 (0.13) | 0.18 (0.13)
Statistical Analysis 1: Comparison: Year 1 Change vs Year 2 Change; Test type: Superiority or Other; p < 0.001, signed rank test

25. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, and Discontinuations Reported During the Double-blind Period
Description: as for outcome 10
Time Frame: Includes data up to 56 days post the last dose in the double-blind period or start of the open-label period, whichever occurred first.
Population: All treated participants in the Double-Blind period
Measure: Number; unit: participants
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 256 | 253
participants
  Deaths | 2 | 4
  SAEs | 20 | 20
  Related SAEs | 5 | 6
  Discontinued due to SAEs | 3 | 3
  AEs | 217 | 211
  Related AEs | 98 | 114
  Discontinued due to AEs | 8 | 11

26. Secondary Outcome: Number of Participants With Laboratory Values Meeting the Marked Abnormality Criteria During the Double-blind Period
Description: Number of participants with laboratory values (hematology, liver and kidney functions, electrolytes, glucose tests, protein tests, metabolite tests, and urine chemistry tests) considered markedly abnormal according to prespecified protocol criteria
Time Frame: as for outcome 25
Population: All treated in the DB period. n=Number of participants evaluated for this measure.
Measure: Number; unit: participants
Arm/Group | ABA + MTX (Double-Blind) | PLA + MTX (Double-Blind)
Number analyzed (Participants) | 256 | 253
participants
  Low Hemoglobin (n=254; n=251) | 3 | 3
  Low Hematocrit (n=254; n=250) | 1 | 2
  Low Erythrocytes (n=254; n=250) | 1 | 4
  Low Platelet Count (n=252; n=250) | 0 | 1
  High Platelet Count (n=252; n=250) | 1 | 3
  Low Leukocytes (n=254; n=251) | 5 | 11
  High Leukocytes (n=254; n=251) | 5 | 14
  Low Neutrophils + Bands (absolute) (n=254; n=252) | 2 | 5
  Low Lymphocytes (absolute) (n=254; n=252) | 13 | 29
  High Lymphocytes (absolute) (n=254; n=252) | 0 | 0
  High Monocytes (absolute) (n=254; n=252) | 1 | 1
  High Basophils (absolute) (n=254; n=252) | 0 | 0
  High Eosinophils (absolute) (n=254; n=252) | 7 | 13
  High Alkaline Phosphatase (n=254; n=253) | 1 | 0
  High Aspartate Aminotransferase (n=254; n=253) | 7 | 14
  High Alanine Aminotransferase (n=254; n=253) | 15 | 21
  G-Glutamyl Transferase (n=254; n=253) | 11 | 9
  High Bilirubin, Total (n=254; n=253) | 0 | 2
  High Blood Urea Nitrogen (n=254; n=253) | 9 | 10
  High Creatinine (n=254; n=251) | 33 | 32
  Low Sodium, Serum (n=254; n=253) | 0 | 1
  High Sodium, Serum (n=254; n=253) | 2 | 0
  Low Potassium, Serum (n=254; n=251) | 6 | 3
  High Potassium, Serum (n=254; n=251) | 3 | 2
  Low Chloride, Serum (n=254; n=253) | 0 | 0
  High Chloride, Serum (n=254; n=253) | 1 | 0
  Low Calcium, Total (n=254; n=253) | 0 | 0
  High Calcium, Total (n=254; n=253) | 0 | 0
  Low Phosphorus, Inorganic (n=254; n=251) | 1 | 2
  High Phosphorus, Inorganic (n=254; n=251) | 3 | 3
  Low Glucose, Serum (n=254; n=253) | 22 | 24
  High Glucose, Serum (n=254; n=253) | 10 | 13
  Low Protein, Total (n=254; n=253) | 2 | 0
  High Protein, Total (n=254; n=253) | 0 | 1
  Low Albumin (n=254; n=253) | 2 | 5
  High Protein, Urine (n=252; n=250) | 6 | 3
  High Glucose, Urine (n=252; n=250) | 4 | 6
  High Blood, Urine (n=252; n=250) | 30 | 22
  High Leukocyte Esterase (n=87; n=88) | 13 | 13
  High Red Blood Cells, Urine (n=92; n=103) | 30 | 25
  High White Blood Cells, Urine (n=94; n=105) | 38 | 42
  High Uric Acid (n=254; n=253) | 1 | 1

ADVERSE EVENTS:
Groups:
- Abatacept: ABA 10 mg/kg (weight-tiered dose) intravenous (IV) infusions in combination with oral MTX titrated to at least 15 mg per week not to exceed 20 mg per week. Study drug administered on Days 1, 15, 29 and every 28 days thereafter up to Month 12.
- Placebo: Placebo (Dextrose 5% Water for Injection U.S.P. [D5W] or Normal Saline [NS] IV infusions in combination with oral MTX titrated to at least 15 mg per week not to exceed 20 mg per week. Administered on Days 1, 15, 29, and every 28 days thereafter up to Month 12.
Arm/Group | Abatacept | Placebo
Serious Adverse Events (participants affected / at risk) | 20/256 | 20/253
Other Adverse Events (participants affected / at risk) | 150/256 | 155/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (N=256) | Placebo (N=253)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 2 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 1
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 3
CELLULITIS (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 1
BREAST CELLULITIS (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 | 0
URETHRAL STENOSIS (Renal and urinary disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CRYPTOGENIC ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SUDDEN DEATH (General disorders) | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 0 | 1
INFUSION RELATED REACTION (General disorders) | 1 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEOPLASM SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (N=256) | Placebo (N=253)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 16 | 13
HYPERTENSION (Vascular disorders) | 17 | 14
HEADACHE (Nervous system disorders) | 30 | 23
DIZZINESS (Nervous system disorders) | 19 | 13
NAUSEA (Gastrointestinal disorders) | 26 | 41
DIARRHOEA (Gastrointestinal disorders) | 17 | 24
DYSPEPSIA (Gastrointestinal disorders) | 11 | 14
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 9 | 15
INFLUENZA (Infections and infestations) | 19 | 23
BRONCHITIS (Infections and infestations) | 18 | 12
NASOPHARYNGITIS (Infections and infestations) | 21 | 26
URINARY TRACT INFECTION (Infections and infestations) | 17 | 22
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 26 | 26
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 | 14
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other